CLINICAL TRIAL: NCT02644980
Title: Target Controlled Infusion of Etomidate or Propofol for Anesthesia of Thoracoscopic Mitral Valve Replacement Surgery,A Randomized Controlled Double-Blinded Study
Brief Title: Target Controlled Infusion of Etomidate or Propofol for Anesthesia of Thoracoscopic Mitral Valve Replacement Surgery
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Xijing Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: XJZH20140722
Record Dates: First submitted 2014-08-18; First posted 2016-01-01 (Estimated); Last update posted 2016-01-01 (Estimated); Status verified 2015-12

CONDITIONS: Delirium; Hemodynamic Instability
Keywords: Target Controlled Infusion
MeSH Terms: conditions — Delirium | interventions — Propofol; Etomidate; Consciousness Monitors; Intubation, Intratracheal

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Etomidate (Experimental): The initiate drug concentration of etomidate is set to 0.2 μg/ml, increasing 0.1 μg/ml every minutes until the BIS(Bispectral index ) reaches 40~60.
  Interventions: Drug: Etomidate; Device: Bispectral Index Monitor; Drug: Induction of anesthesia; Drug: Maintenance of anesthesia; Other: Tracheal Intubation
- Propofol (Experimental): The initiate drug concentration of propofol is set to 1.0 μg/ml, increasing 0.3 μg/ml every minutes until the BIS(Bispectral index ) reaches 40~60.
  Interventions: Drug: Propofol; Device: Bispectral Index Monitor; Drug: Induction of anesthesia; Drug: Maintenance of anesthesia; Other: Tracheal Intubation

INTERVENTIONS:
Drug: Propofol — The initiate drug concentration of propofol is set to 1.0 μg/ml, increasing 0.3 μg/ml every minutes until the BIS(Bispectral index ) reaches 40~60.
  Arms: Propofol
Drug: Etomidate — The initiate drug concentration of etomidate is set to 0.2 μg/ml, increasing 0.1 μg/ml every minutes until the BIS(Bispectral index ) reaches 40~60.
  Other Names: Fuerli
  Arms: Etomidate
Device: Bispectral Index Monitor — BIS monitored from beginning of anesthesia induction to the end of the surgery.
  Other Names: BIS
Drug: Induction of anesthesia — Midazolam 0.03 mg/kg injection vein，Sufentanyl 0.5~1 μg/kg, target controlled infusion of etomidate or propofol,after the consciousness of patients is lost, rocuronium 0.6mg/kg is given.
Drug: Maintenance of anesthesia — After the intubation, target controlled infusion(TCI) of etomidate or propofol is maintained,rocuronium 0.15mg/kg and sufentanil is given when needed. When the operation is over, the TCI is stopped.
Other: Tracheal Intubation — After the induction of anesthesia, Tracheal intubation is performed.

SUMMARY:
For patients requiring the heart valve replacement surgery, heart function is injured in different degree.Thus, minimizing the impact of the anesthesia drug on the cardiovascular system has important clinical meanings. Etomidate has slight effect on the cardiovascular system, often used in the induction of anesthesia, however target controlled infusion etomidate in maintenance of anesthesia is less used. So, the trial is designed to observe the application value of TCI etomidate in thoracoscopic mitral valve replacement surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18~75 years old
2. Selective cardiopulmonary bypass thoracoscopic mitral vales replacement surgery
3. Received heart surgery for the first time
4. New York Heart Association(NYHA) II~III
5. Written informed consent -

Exclusion Criteria:

1. Emergency surgery
2. Anticipated survival time <1 yrs
3. Serious heart, brain, liver,kidney,lung,endocrine diseases or serious infection
4. Prolonged use of hormone or history of adrenal suppression disease
5. Severe mediastinal fiber thickening or fibrous adhesions
6. Allergy to experimental drug or other contraindications
7. Occurred or expected occurring of difficulty airway
8. Sure or suspected narcotic analgesics abuse
9. History of neuro-muscular disease
10. Mental instability or metal disease
11. Pregnancy or brest-feeding
12. Participated other clinical trial past 30 days
13. Malignant hyperthermia

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2015-12; Primary Completion 2016-08 (Estimated); Study Completion 2016-08 (Estimated)

PRIMARY OUTCOMES:
Blood pressure | from the beginning of induction to the surgery over, up to 6 hrs.
  blood pressure(systolic blood pressure and diastolic blood pressure) is monitored and recorded at 9 time points, including 10 minutes before induction,the right moment after induction of anesthesia and tracheal intubation,the beginning of surgery and the cardiopulmonary bypass(CPB),the time the ascending aorta is blocked and unstuck,the time the CPB and the surgery is over.

SECONDARY OUTCOMES:
Heart rate | from the beginning of induction to the surgery over, up to 6 hrs.
  Heart rate is monitored and recorded at 9 time points, including 10 minutes before induction,the right moment after induction of anesthesia and tracheal intubation,the beginning of surgery and the cardiopulmonary bypass(CPB),the time the ascending aorta is blocked and unstuck,the time the CPB and the surgery is over.
Delirium | The right moment of patients'leaving off PACU, expected to be 2 h from the end the of operation
  Using Confusion Assessment Method for the Intensive Care Unit(CAM-ICU) to screening of delirium.
Life quality | at the time of one month right after the surgery
  using the Activities of Daily Living (ADL) to assess the life quality one month after the surgery.
Number of Participants with Serious and Non-Serious Adverse Events | Up to 1 month
  Number of Participants with Serious and Non-Serious Adverse Events including major adverse cardiovascular and cerebrovascular event such as cardiac infraction,stroke, acute renal failure, re-surgery,and death.
  Safety Issue?: Yes
Time of recovery from anesthesia | from the time TCI is stopped to the time patients' eyes open after the surgery, up to 30 minutes.
Bispectral index (BIS) value | from the beginning of induction to the surgery over, up to 6 hrs.
  BIS is monitored and recorded at 9 time points, including 10 minutes before induction,the right moment after induction of anesthesia and tracheal intubation,the beginning of surgery and the cardiopulmonary bypass(CPB),the time the ascending aorta is blocked and unstuck,the time the CPB and the surgery is over.
onset time | The time from TCI etomidate or propofol to the disappearance of eyelash reflex,up to 10 minutes.
  The time period from TCI etomidate or propofol to the disappearance of eyelash reflex.

OTHER OUTCOMES:
Respiratory rates(HR) | from the beginning of induction to the surgery over, up to 6 hrs.
  Respiratory rate is monitored and recorded at 9 time points, including 10 minutes before induction,the right moment after induction of anesthesia and tracheal intubation,the beginning of surgery and the cardiopulmonary bypass(CPB),the time the ascending aorta is blocked and unstuck,the time the CPB and the surgery is over.
pulse blood oxygen saturation (SPO2) | from the beginning of induction to the surgery over, up to 6 hrs.
  pulse blood oxygen saturation is monitored and recorded at 9 time points, including 10 minutes before induction,the right moment after induction of anesthesia and tracheal intubation,the beginning of surgery and the cardiopulmonary bypass(CPB),the time the ascending aorta is blocked and unstuck,the time the CPB and the surgery is over.
Dosage of anesthesia drug | from the beginning of induction of anesthesia to the surgery over, up to 6 hrs.
  record the dosage of the anesthesia drug including propofol and etomidate, sufentanyl and rocuronium used during the period of maintenance of anesthesia.